CLINICAL TRIAL: NCT06446037
Title: Assessment of Gesture Accuracy for a Multi-electrode EMG Sensor Array Based Prosthesis Control System
Brief Title: Assessment of Gesture Accuracy of a Prosthesis Control System
Acronym: ASCENT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Phantom Neuro Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PN01
Record Dates: First submitted 2024-05-28; First posted 2024-06-06 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Upper Limb Amputation Below Elbow (Injury)
Keywords: Prosthesis; Upper limb amputee
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional arm (Experimental): All subjects will be instrumented with an electrode array on their forearms. The EMG signals detected by the electrodes will be fed into Phantom X hardware running the Phantom X algorithms. The algorithms will decode the EMGs signals and drive a desk mounted hand prosthesis.
  Interventions: Device: Non-invasive EMG band instrumentation

INTERVENTIONS:
Device: Non-invasive EMG band instrumentation — The sensed EMG signals from the subjects will be decoded by Phantom X algorithm and used to drive various gestures in a desk-mounted hand prosthesis
  Other Names: EMG prosthesis control

SUMMARY:
The study is evaluating the performance of prosthesis control system, referred to as Phantom X, in able bodied individuals and individuals with upper limb amputation at the forearm level.

DETAILED DESCRIPTION:
The study will characterize the performance of Phantom X system and associated algorithms in decoding EMG signals for various hand gesture control. The EMG signals will be sensed using a non-invasive multi-electrode array applied to subjects' forearms.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 21 years in age and older
2. Individuals with amputation of one or both arms at transradial level (applies to amputees only)
3. Ability to follow study directions
4. Willingness and ability to sign Informed Consent

Exclusion Criteria:

1. Individuals with previously diagnosed muscle pathologies
2. Individuals with impaired muscle function and/or impaired ability to perform normal hand movements (normal participants) or ability to perform normal phantom hand movements (amputees)
3. Individuals with transhumeral or higher amputation of both arms (applies to amputees only)
4. Cognitively impaired to follow study instructions
5. Allergies to skin adhesive materials necessary for cutaneous electrode placement
6. Excessive hair growth on arms and inability to shave off the hair for electrode placement
7. Pregnant woman
8. Arms or residual limbs with insufficient diameter to accommodate the wearing of two cutaneous sensor arrays
9. Injuries, bruises, or open wounds on the arm that needs to be instrumented for the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Gesture accuracy | Acute visit (at most 3 hours)
  Percentage of hand gestures accurately decoded by Phantom X algorithm

CONTACTS AND LOCATIONS:
Locations (1):
- Phantom Neuro Inc. Operational Headquarters, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No